CLINICAL TRIAL: NCT06448819
Title: Real-life Use of the Crohn's Disease Exclusion Diet (CDED) in Adult Patients With Mild-to-moderate Crohn's Disease Activity: an Open Label, Randomized Controlled Trial
Brief Title: Real-life Use of the Crohn's Disease Exclusion Diet (CDED) in Adult Patients With Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Giorgia Bodini, Prof, Universita degli Studi di Genova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDED-1
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDED group (Experimental): Crohn's disease exclusion diet Partecipants received Crohn's disease exclusion diet or Mediterranean diet for 24 weeks
  Interventions: Other: Diet
- Mediterranean group (No Intervention)

INTERVENTIONS:
Other: Diet — Patients received Crohn's disease exclusion diet or Mediterranean diet
  Arms: CDED group

SUMMARY:
This study explores the effectiveness od the Crohn's Disease Exclusion Diet (CDED) as a tretament for adults with mild-to-moderate Crohn's disease (CD). The hypotesis is that CDED, by excluding specific dietary components thought to exacerbate gut inflammation, can induce remission in CD patients more effectively than a control diet based on the Mediterranean pattern. Conducted as an open-label randomized trial, the research aim to provide real-world evidence of CDED's safety and its inpact on clinical remission, body composition and overall quality of life for CD patients.

ELIGIBILITY:
Inclusion Criteria:

* mild-to-moderate Crohn's disease activity (HBI between 5 and 16)

Exclusion Criteria:

* concomitant treatment with corticosteroids, antibiotic therapies and nutraceutical supplements, treatment with biological drugs and traditional immunosuppressants started less than 24 weeks before enrollment, presence of active fistulas or abscesses, gastrointestinal tract surgery less than 6 months to randomization, coeliac disease, type 1 diabetes mellitus, uncontrolled type 2 diabetes mellitus, acute coronary disease (unstable angina, myocardial infarction), advanced acute or chronic liver disease, congestive heart failure (NYHA class III-IV), acute and chronic nephropathies (GRF<30 ml/min according to the CKD-EPI formula), presence of acute infectious diseases and pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Harvey-Bradshaw Index (HBI | 12 weeks; 24 weeks

SECONDARY OUTCOMES:
Fecal calprotectin | 12 weeks; 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Giorgia Bodini, Genova, Italy

IPD SHARING:
Plan to Share IPD: No